CLINICAL TRIAL: NCT04165109
Title: Alzheimer's Clinical Trial Consortium for Down Syndrome (ACTC-DS) Trial-Ready Cohort - Down Syndrome (TRC-DS)
Brief Title: Trial-Ready Cohort-Down Syndrome (TRC-DS)
Acronym: TRC-DS
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Clinical Trials Consortium (Other); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Michael Rafii, MD, PhD, Professor, University of Southern California
Other Study IDs: ATRI-006; 1R61AG066543-01 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-11-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome; Alzheimer Disease; Dementia
Keywords: Trial-Ready Cohort; Observational; Alzheimer's; Prevention; Down Syndrome
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trial Ready Cohort: Non-demented adults with Down syndrome (DS)

SUMMARY:
The purpose of the Trial-Ready Cohort - Down Syndrome (TRC-DS) is to enroll 120 healthy adults with Down syndrome (DS), between the ages of 25-55, into a trial ready cohort (TRC), and up to 450 participants in total including co-enrolled in the Alzheimer Biomarkers Consortium - Down Syndrome (ABC-DS) study. Participants enrolled in the TRC-DS will undergo longitudinal cognitive and clinical assessment, genetic and biomarker testing, as well as imaging and biospecimen collection. Using these outcome measures, researchers will analyze the relationships between cognitive measures and biomarkers of Alzheimer's disease (AD) to identify endpoints for AD clinical trials in DS that best reflect disease progression.

To learn more about the study and participating sites, visit our study website at: https://www.trcds.org/.

TRC-DS is collaborating with the Alzheimer's Disease Biomarker Consortium-Down Syndrome (ABC-DS) to allow study participants to be concurrently enrolled in both ABC-DS and TRC-DS, referred to as "co-enrollment". ABC-DS is a longitudinal, observational research study that is overseen at University of Pittsburgh Coordinating Center. ABC-DS participants who express interest in potentially joining a clinical trial in the future and who meet TRC-DS eligibility criteria, may choose to co-enroll in TRC-DS at an ABC-DS Site. Co-enrolled participants will adhere to the ABC-DS protocol and schedule of activities, but agree to share their data with the TRC-DS team and to receive invitations for future participation in clinical trials. Fore more information on ABC-DS please visit https://www.nia.nih.gov/research/abc-ds or http://abcds.pitt.edu/.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DS (including trisomy 21, mosaic trisomy 21, Robertsonian translocation trisomy 21 or partial trisomy 21) (as confirmed by Karyotype genetic testing or medical record review)
2. Provision of signed and dated informed consent form; this includes adults with DS who can provide consent, or for whom an LAR provides consent on behalf of the individual to participate. Adults with DS who cannot consent must sign and date an assent accompanied with a signed and dated consent by legally authorized representative (LAR).
3. Stated availability and willingness to comply with all study procedures and availability for the duration of the study or until referred to a clinical trial
4. Male or female, aged 25-55 inclusive
5. In good general health as evidenced by medical history with no diagnosis of dementia
6. Permitted CNS-active medications, stable in dose for at least 4 weeks or longer. If new medications have been started, medical monitoring team will review on case by case basis to recommend timing of baseline cognitive testing
7. Adequate visual and auditory acuity to allow neuropsychological testing
8. Mental Age of 4 years or greater (based upon the Kaufman Brief Intelligence Test, Second Edition, or based upon medical records)
9. IQ equal to or greater than 40 (based upon the Kaufman Brief Intelligence Test, Second Edition)
10. Must speak English or Spanish fluently
11. Must have a reliable Study Partner (may be caregiver, sibling, parent) who is capable of providing correct information about the participant's clinical symptoms and history

Exclusion Criteria:

1. Any significant disease or unstable medical condition that could affect participation (i.e., unstable psychiatric disease, unstable cardiac problems, chronic renal failure, chronic hepatic disease, severe pulmonary disease)
2. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant (Dental fillings do not present a risk for MRI)
3. Participants unable to complete MRI procedure
4. History, within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
5. Clinically significant abnormalities in B12 or TFTs that might interfere with the study. A low B12 is exclusionary, unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant. A high TSH is exclusionary unless follow up T3/T4 levels indicate that it is not physiologically significant.
6. Clinically significant abnormalities in screening laboratories
7. For participants undergoing CSF collection: a current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening or if on anti-coagulation therapy (e.g. warfarin)
8. Concurrent participation in a clinical trial for an investigational product or concurrent participation in longitudinal study with overlapping outcome measures/procedures is prohibited with the exception of ABC-DS co-enrollment or as approved by project director
9. Participants whom the investigator deems to be otherwise ineligible. The Investigators should consult with the Coordinating Center on any issues that may disqualify the participant from participation in future clinical trials to determine whether enrollment into TRC-DS would be appropriate

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 120 non-demented adults with Down Syndrome and up to 450 participants in total including co-enrollment the Alzheimer Biomarkers Consortium - Down Syndrome (ABC-DS)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment of participants into the Trial-Ready Cohort in DS (TRC-DS). | 5 years
  The primary aim of the TRC-DS is enrollment of 120 participants into the trial ready cohort, with up to 450 participants in total including co-enrollment with the Alzheimer Biomarkers Consortium - Down Syndrome (ABC-DS) study, to support future referral and enrollment into primary Alzheimer's disease (AD) prevention trials for adults with DS.

SECONDARY OUTCOMES:
Change in cognition as measured by the Cued Recall Test | Baseline and Month 32, or until enrollment into a clinical trial
  The Cued Recall Test is modified from a version developed for adults from the typical population. Twelve items are presented for learning, 4 at a time, with each item accompanied by a unique category cue. The testing phase consists of 3 trials. Each trial begins with free recall of the test items; following free recall, a category cue is provided for those items not spontaneously recalled. Two scores are generated from the test, a Free Recall Score and a Total Score (Free Recall plus items recalled when the category cue is provided). A cut-off of < 23 on the Total Score resulted in a sensitivity of 91% and a specificity of 84% when individuals with DS and a diagnosis of dementia were compared to their healthy peers without dementia.
Change in behavior as measured by the Neuropsychiatric Inventory (NPI) | Screening and Month 32, or until enrollment into a clinical trial
  The Neuropsychiatric Inventory (NPI) is a well-validated, reliable, multi-item instrument to assess psychopathology in AD based on an interview with a caregiver or qualified study partner. It evaluates both the frequency and severity of 12 neuropsychiatric features including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, and appetite and eating disorders. A higher NPI score means that the participant is displaying more behavioral symptoms. The minimum score is 0 and the maximum is 144. A score of 0-20 is mild, 20-50 moderate and greater than 50 means significant behavioral symptoms.
Change in cognition as measured by the Down Syndrome Mental Status Exam (DSMSE) | Screening and Month 32, or until enrollment into a clinical trial
  The DSMSE is an omnibus measure of neuropsychological function that assesses a broad range of skills and is easy to administer. It is divided into items that test recall for personal information, orientation to season and day of week, memory, language, visuospatial function, and praxis. Recall for personal information is tested with questions about the subject's name, age and birth date. Orientation items ask the day of the week and season of the year. Memory in the DSMSE is assessed with items that require immediate and delayed recall of three objects and for the location of three hidden objects. Language items include confrontation naming, sentence repetition, and comprehension of one, two, and three step commands. Visuospatial items are three-dimensional block constructions. Praxis items include transitive and intransitive limb movements and a sequential task.
Change in behavior as measured by the Vineland 3 (Informant Version) | Baseline and Month 32, or until enrollment into a clinical trial
  The Vineland Adaptive Behavior Scale 3 (VABS-II) I is a normed assessment tool that assesses adaptive behavior across the areas of communication, activities of daily living, and socialization. The tool is self-administered via interview toby a study partner using a tablet (e.g. iPad), takes approximately 45 minutes to complete and may be done remotely.
  The VABS-III scores range from 20-140. Higher scores indicate higher functioning. Specifically, these include 'very high' (domain and Adaptive Behavior Scale (ABC) Standard Scores of 130-140), "moderately high" (domain and ABC Standard Scores of 115-129), "adequate" (domain and ABC Standard Scores of 86-114), "moderately low" (domain and ABC Standard Scores of 71-85), and "low" (domain and ABC Standard Scores of 20-70).
Change in cognition as measured by the National Task Group Early Detection Screen for Dementia (NTG-EDSD) | Baseline and Month 32, or until enrollment into a clinical trial
  The National Task Group Early Detection Screen for Dementia (NTG-EDSD) is a screening tool which measures changes typically observed in dementia. It is composed of four primary sections about relative demographics, ratings of health, mental health, and life stressors, a review of multiple domains associated with adult functioning, and a review of chronic medical conditions. The NTG-EDSD is completed by a staff member who interviews the caregiver. It contains 40 questions/question groups and takes 15 mins to administer.
Change in cognition as measured by the Stroop Dog and Cat Task | Baseline and Month 32, or until enrollment into a clinical trial
  In the Stroop Dog and Cat Task, a linear sequence of 16 pictures (8 cats, 8 dogs) are presented in a pre-determined random order. In the control condition the subject says the name of each picture and is urged to do so rapidly. In the experimental (inhibition) condition the participant is required to say 'cat' for the picture of each dog and 'dog' for the cat. For each condition the participant is given a brief practice period. Performance on the Stroop Dog and Cat was significantly related to informant-reported memory changes in 103 adults with DS with mild-moderate intellectual disability in the age range of 36 - 72 years.
Change in brain volume as measured by magnetic resonance imaging (MRI) | Baseline and Month 32, or until enrollment into a clinical trial
Change in plasma Amyloid Beta (Abeta) biomarkers | Baseline and Month 32, or until enrollment into a clinical trial
Change in plasma tau biomarkers | Baseline and Month 32, or until enrollment into a clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rafii, MD, PhD, Principal Investigator — USC Alzheimer's Therapeutic Research Institute (ATRI)
Locations (20):
- United States (16):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, Irvine School of Medicine, Co-Enrolling through ABC-DS Only, Orange, California
  - Linda Crnic Institute for Down Syndrome, University of Colorado, Aurora, Colorado
  - Advocate Medical Group Adult Down Syndrome Center, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Co-Enrolling through ABC-DS Only, Lexington, Kentucky
  - Massachusetts General Hospital, Co-Enrolling through ABC-DS Only, Boston, Massachusetts
  - Washington University, St. Louis, St Louis, Missouri
  - New York State Institute for Basic Research in Developmental Disabilities (SIBRDD), Co-Enrolling through ABC-DS Only, Staten Island, New York
  - Case Western Reserve University, Beachwood, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Co-Enrolling through ABC-DS Only, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center Center for Cognitive Medicine, Nashville, Tennessee
  - University of Texas Health San Antonio, Glenn Biggs Institute for Alzheimer's & Neurodegenerative Diseases, San Antonio, Texas
  - University of Wisconsin - Madison, Waisman Center, Co-Enrolling through ABC-DS Only, Madison, Wisconsin
- Institut Jerome Lejeune, Paris, France, France
- Institute of Memory & Cognition, Tallaght University Hospital, Dublin, Ireland, Ireland
- Sant Pau Biomedical Research Institute (IIB Sant Pau), Barcelona, Spain
- University of Cambridge, Co-Enrolling through ABC-DS Only, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy J. The discovery of Alzheimer-causing mutations in the APP gene and the formulation of the "amyloid cascade hypothesis". FEBS J. 2017 Apr;284(7):1040-1044. doi: 10.1111/febs.14004. PMID 28054745
- [Background] Selkoe DJ, Hardy J. The amyloid hypothesis of Alzheimer's disease at 25 years. EMBO Mol Med. 2016 Jun 1;8(6):595-608. doi: 10.15252/emmm.201606210. Print 2016 Jun. PMID 27025652
- [Background] Handen BL, Cohen AD, Channamalappa U, Bulova P, Cannon SA, Cohen WI, Mathis CA, Price JC, Klunk WE. Imaging brain amyloid in nondemented young adults with Down syndrome using Pittsburgh compound B. Alzheimers Dement. 2012 Nov;8(6):496-501. doi: 10.1016/j.jalz.2011.09.229. PMID 23102120
- [Background] Rafii MS, Wishnek H, Brewer JB, Donohue MC, Ness S, Mobley WC, Aisen PS, Rissman RA. The down syndrome biomarker initiative (DSBI) pilot: proof of concept for deep phenotyping of Alzheimer's disease biomarkers in down syndrome. Front Behav Neurosci. 2015 Sep 14;9:239. doi: 10.3389/fnbeh.2015.00239. eCollection 2015. PMID 26441570
- [Background] Lao PJ, Betthauser TJ, Hillmer AT, Price JC, Klunk WE, Mihaila I, Higgins AT, Bulova PD, Hartley SL, Hardison R, Tumuluru RV, Murali D, Mathis CA, Cohen AD, Barnhart TE, Devenny DA, Mailick MR, Johnson SC, Handen BL, Christian BT. The effects of normal aging on amyloid-beta deposition in nondemented adults with Down syndrome as imaged by carbon 11-labeled Pittsburgh compound B. Alzheimers Dement. 2016 Apr;12(4):380-90. doi: 10.1016/j.jalz.2015.05.013. Epub 2015 Jun 13. PMID 26079411
- [Background] Rafii MS, Lukic AS, Andrews RD, Brewer J, Rissman RA, Strother SC, Wernick MN, Pennington C, Mobley WC, Ness S, Matthews DC; Down Syndrome Biomarker Initiative and the Alzheimer's Disease Neuroimaging Initiative. PET Imaging of Tau Pathology and Relationship to Amyloid, Longitudinal MRI, and Cognitive Change in Down Syndrome: Results from the Down Syndrome Biomarker Initiative (DSBI). J Alzheimers Dis. 2017;60(2):439-450. doi: 10.3233/JAD-170390. PMID 28946567
- [Background] McCarron M, McCallion P, Reilly E, Dunne P, Carroll R, Mulryan N. A prospective 20-year longitudinal follow-up of dementia in persons with Down syndrome. J Intellect Disabil Res. 2017 Sep;61(9):843-852. doi: 10.1111/jir.12390. Epub 2017 Jun 29. PMID 28664561
- [Background] Firth NC, Startin CM, Hithersay R, Hamburg S, Wijeratne PA, Mok KY, Hardy J, Alexander DC; LonDownS Consortium; Strydom A. Aging related cognitive changes associated with Alzheimer's disease in Down syndrome. Ann Clin Transl Neurol. 2018 May 20;5(6):741-751. doi: 10.1002/acn3.571. eCollection 2018 Jun. PMID 29928657
- [Background] Startin CM, Hamburg S, Hithersay R, Al-Janabi T, Mok KY, Hardy J; LonDownS Consortium; Strydom A. Cognitive markers of preclinical and prodromal Alzheimer's disease in Down syndrome. Alzheimers Dement. 2019 Feb;15(2):245-257. doi: 10.1016/j.jalz.2018.08.009. Epub 2018 Nov 28. PMID 30503169
- [Background] Hithersay R, Startin CM, Hamburg S, Mok KY, Hardy J, Fisher EMC, Tybulewicz VLJ, Nizetic D, Strydom A. Association of Dementia With Mortality Among Adults With Down Syndrome Older Than 35 Years. JAMA Neurol. 2019 Feb 1;76(2):152-160. doi: 10.1001/jamaneurol.2018.3616. PMID 30452522
- See also: ATRI Studies — https://keck.usc.edu/atri/research/studies/
- See also: Alzheimer's Clinical Trials Consortium — https://www.actcinfo.org/
- See also: The INCLUDE Project — https://www.nih.gov/include-project
- See also: Alzheimer's Clinical Trials Consortium - Down syndrome — http://www.actc-ds.org
- See also: Trial Ready Cohort-Down Syndrome — https://www.trcds.org/